CLINICAL TRIAL: NCT04527458
Title: Case Fatalities in Hospitalised COVID-19 Patients in the UK: An ISARIC Study
Brief Title: Case Fatalities in Hospitalised COVID-19 Patients in the UK
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: International Severe Acute Respiratory and Emerging Infection Consortium (Other); BREATHE Health Data Research Hub (Unknown)
Responsible Party: Sponsor
Other Study IDs: ISARIC_COVID_CF
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: COVID-19; ISARIC; Hospitalisations; Mortality; Case fatality; United Kingdom
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Drug Treatment; Triage; Surge Capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalisations: All hospitalised COVID patients
  Interventions: Other: Patient Characteristics; Other: COVID-19 treatments; Other: Differences in triage; Other: Surge capacity
- Critical care: All hospitalised COVID patients in critical care
  Interventions: Other: Patient Characteristics; Other: COVID-19 treatments; Other: Differences in triage; Other: Surge capacity

INTERVENTIONS:
Other: Patient Characteristics — Characteristics of the patients
Other: COVID-19 treatments — Specific treatments used on COVID-19 patients
Other: Differences in triage — Triage criteria for treating COVID-19 patients
Other: Surge capacity — Capacity of hospitals

SUMMARY:
This study will investigate how the case fatality in hospitalised patients with COVID-19 has changed throughout the pandemic. It will also explore possible mechanisms that could be driving these changes. This analysis will enhance our understanding of the virus, which will be important for researchers and clinicians to respond appropriately.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted with a proven or high likelihood of COVID-19

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with proven or high likelihood of COVID-19 admitted to the 260 UK hospitals enrolled in the ISARIC-4C study
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2020-08-02 (Actual)

PRIMARY OUTCOMES:
Case fatality | 23 weeks
  The proportion of new admissions with COVID-19 who died over time

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie B Docherty, Principal Investigator — Usher Institute, University of Edinburgh; Ewen M Harrison, Principal Investigator — Usher Institute, University of Edinburgh; Rachel H Mulholland, Principal Investigator — Usher Institute, University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to all data and samples collected by ISARIC4C are controlled by an Independent Data and Materials Access Committee (IDAMAC), composed of representatives of research funders, academia, clinical medicine, public health and industry. Their job is to ensure that all data and samples are used to generate the greatest possible benefit to humanity, in the shortest possible time.

REFERENCES:
- [Background] Docherty AB, Harrison EM, Green CA, Hardwick HE, Pius R, Norman L, Holden KA, Read JM, Dondelinger F, Carson G, Merson L, Lee J, Plotkin D, Sigfrid L, Halpin S, Jackson C, Gamble C, Horby PW, Nguyen-Van-Tam JS, Ho A, Russell CD, Dunning J, Openshaw PJ, Baillie JK, Semple MG; ISARIC4C investigators. Features of 20 133 UK patients in hospital with covid-19 using the ISARIC WHO Clinical Characterisation Protocol: prospective observational cohort study. BMJ. 2020 May 22;369:m1985. doi: 10.1136/bmj.m1985. PMID 32444460
- See also: ISARIC 4C website — https://isaric4c.net/